CLINICAL TRIAL: NCT04776486
Title: Evaluation of Glomerular Filtration Rate Using Iohexol Plasma Clearance in Critically Ill Patients With Augmented Renal Creatinine Clearance
Brief Title: Iohexol Clearance in Critically Ill Patients With Augmented Renal Creatinine Clearance
Acronym: GFR-ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190414; 2019-A00654-53 (Other: IDRCB)
Record Dates: First submitted 2020-07-17; First posted 2021-03-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Augmented Renal Clearance; Critically Ill
Keywords: Iohexol; Augmented renal clearance; Intensive Care Unit
MeSH Terms: conditions — Critical Illness | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Critically ill patients with augmented renal clearance (Experimental): ICU patients with estimated renal clearance over 130ml/min/1.73m2
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Iohexol — Intravenous injection of 5 ml of iohexol (Omnipaque) to calculate the glomerular filtration rate (area under the curve).
  Blood samples (2 ml) and urine (2 ml minimum) are to be collected for the determination of iohexol clearance at the following time points: pre-dose, 5 minutes, and 1, 2, 3, 4, 5, 6 hours post dose.
  Other Names: Omnipaque

SUMMARY:
Evaluation of glomerular filtration rate using iohexol plasma clearance in critically ill patients with augmented renal creatinine clearance

DETAILED DESCRIPTION:
Single center study in ICU patients with augmented renal clearance comparing glomerular filtration rate (GFR) as measured by iohexol plasma clearance to that measured by creatinine clearance. Primary objective is to compare the GFR estimates made by iohexol plasma clearance (as reference method) and creatinine clearance using Bland-Altman method.

Secondary objective are to compare GFR as measured by iohexol plasma clearance to that calculated with the most commonly used renal clearance estimating formulas (Cockcroft and Gault, MDRD and CKD-EPI ), evaluate clinical determinant of the observed differences and evaluate determinants of extracellular volume.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient
* 24h Creatinine clearance >130ml/min/1.73m2
* Urinary catheterization
* Affiliation to a social security scheme

Exclusion Criteria:

* Pregnancy
* CT-scan with contrast media infusion the day of inclusion
* Documented allergy to contrast media
* Patient under guardianship / curatorship
* Patient benefiting from the "State Medical Assistance"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2026-01-29 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
GFR obtained by the iohexol clearance technique | 6 hours
  GFR as measured by iohexol plasma clearance to evaluate its concordance, by the Bland and Altman method, with that obtained by measuring the clearance of creatinine.
GFR obtained by the creatinine clearance technique | 6 hours
  GFR as measured by creatinine plasma clearance

SECONDARY OUTCOMES:
GFR calculated using the Cockroft-Gault equation | 6 hours
  Estimation of GFR using the Cockroft-Gault method based on the serum creatinine clearance measured on the day of intervention and the patient's weight of the day, and the agreement with the GFR measured by the iohexol clearance
GFR calculated using the Modification of diet in renal disease (MDRD) formula | 6 hours
  Estimation of GFR using MDRD method based on the serum creatinine clearance measured on the day of intervention and the patient's weight of the day, and the agreement with the GFR measured by the iohexol clearance
GFR calculated using the Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI) equation | 6 hours
  Estimation of GFR using CKD-EPI method based on the serum creatinine clearance measured on the day of intervention and the patient's weight of the day, and the agreement with the GFR measured by the iohexol clearance
Plasmatic Levetiracetam dosing | 6 hours
  To detect underdosing and risk of therapeutic failure of Levetiracetam
Plasmatic Vancomycin dosing | 6 hours
  To detect underdosing and risk of therapeutic failure of Vancomycin
Plasmatic Piperacillin dosing | 6 hours
  To detect underdosing and risk of therapeutic failure of Piperacillin
Plasmatic Cefotaxim dosing | 6 hours
  To detect underdosing and risk of therapeutic failure of Cefotaxim
Plasmatic Aminoglycoside dosing | 6 hours
  To detect underdosing and risk of therapeutic failure of Aminoglycoside

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin G Chousterman, MD PhD, Principal Investigator — Lariboisière Hospital, APHP Nord
Locations (1):
- Lariboisière Hospital, Surgical ICU, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salmon-Gandonniere C, Benz-de Bretagne I, Mercier E, Joret A, Halimi JM, Ehrmann S, Barin-Le Guellec C. Iohexol clearance in unstable critically ill patients: a tool to assess glomerular filtration rate. Clin Chem Lab Med. 2016 Nov 1;54(11):1777-1786. doi: 10.1515/cclm-2015-1202. PMID 27166722